CLINICAL TRIAL: NCT04414228
Title: An Investigation of the Impact of Anesthetic Guidance of Depth of Anesthesia and Indirect Cardiac Output Monitoring on the Clinical Outcomes of Patients Undergoing Thoracic Surgery: A Factorial Parallel Randomized Controlled Trial
Brief Title: Anesthetic Guidance of Depth of Anesthesia and Indirect Cardiac Output Monitoring in Thoracic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Principal Investigator, YingHsuanTai, Department of Anesthesiology, Taipei Medical University Shuang Ho Hospital
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: N202004045
Record Dates: First submitted 2020-05-29; First posted 2020-06-04 (Actual); Last update posted 2022-05-18 (Actual); Status verified 2022-05

CONDITIONS: Anesthesia; Hemodynamic Instability; Postoperative Respiratory Complication

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- M-Entropy guidance of anesthesia depth (Active Comparator): In the M-Entropy group, dosage of volatile anesthetics will be adjusted to achieve the response and state entropy values between 40 and 60 from the start of anesthesia to the end of surgery. In the control group, dosage of volatile anesthetics will be titrated according to clinical judgment.
  Interventions: Device: M-Entropy guidance of anesthesia depth
- ProAQT in guiding goal-directed hemodynamic therapy (Active Comparator): Subjects randomized to the GDT group will be managed according to the ERAS algorithm utilizing ProAQT variables (mean arterial pressure, stroke volume variation and cardiac index) If stroke volume variation is ≥ 10%, a bolus of 150 ml of crystalloid fluid will be given until the stroke volume variation is < 10%. If mean arterial pressure is < 70 mmHg and/or cardiac index < 2.5 l·min-1·m-2 despite the stroke volume variation of < 10% following fluid challenge, single or consecutive boluses of ephedrine 4 mg and/or continuous intravenous infusion of norepinephrine 2-10 μg·min-1 will be administered.
  Interventions: Device: ProAQT in guiding goal-directed hemodynamic therapy

INTERVENTIONS:
Device: M-Entropy guidance of anesthesia depth — In the M-Entropy group, dosage of volatile anesthetics will be adjusted to achieve the response and state entropy values between 40 and 60 from the start of anesthesia to the end of surgery. In the control group, dosage of volatile anesthetics will be titrated according to clinical judgment.
  Arms: M-Entropy guidance of anesthesia depth
Device: ProAQT in guiding goal-directed hemodynamic therapy — If stroke volume variation is ≥ 10%, a bolus of 150 ml of crystalloid fluid will be given until the stroke volume variation is < 10%. If mean arterial pressure is < 70 mmHg and/or cardiac index < 2.5 l·min-1·m-2 despite the stroke volume variation of < 10% following fluid challenge, single or consecutive boluses of ephedrine 4 mg and/or continuous intravenous infusion of norepinephrine 2-10 μg·min-1 will be administered.
  Arms: ProAQT in guiding goal-directed hemodynamic therapy

SUMMARY:
Patients undergoing thoracotomy in thoracic surgery are prone to have complications of delayed recovery from general anesthesia and perioperative instable hemodynamics due to the relatively invasive procedures and patient's underlying morbidity. Therefore, intraoperative monitoring and corresponding management are of great importance to prevent relevant complications in thoracic surgery. This study aims to investigate the clinical benefits of two intraoperative monitoring techniques in patients undergoing thoracotomy surgery, including depth of anesthesia and minimally invasive cardiac output monitoring. First, M-Entropy system will be used to measure the depth of anesthesia and be evaluated regarding the effect of spectral entropy guidance on postoperative recovery. Second, we will apply ProAQT device in guiding goal-directed hemodynamic therapy and assess its impact on occurrence of postoperative pulmonary complications and recovery. In this study, we will conduct a factorial parallel randomized controlled trial and use the method of stratified randomization to evaluate both two monitoring technologies in the same patient group. The results of this study will provide important evidence and clinical implication for precision anesthesia and enhanced recovery after surgery (ERAS) protocol in thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing video-assisted thoracotomy for lung resection at Shuang Ho Hospital, Taipei Medical University, New Taipei City, Taiwan.

Exclusion Criteria:

* Age < 20 years
* Pregnancy
* End-stage renal disease
* Emergency surgery
* Presence of circulatory shock needing vasoactive drugs before surgery
* Any diagnosis of aortic diseases
* Cerebral vascular diseases or trauma
* High-degree cardiac arrythmia (e.g. atrial fibrillation)
* Uses of cardiac pacemaker or automated implantable cardioverter defibrillator
* New York Heart Association functional classification 4
* Long-term use of psychiatric medications
* Intraoperative blood loss > 1 L
* Intraoperative blood transfusion
* Planned or unanticipated transferal to ICU for postoperative mechanical ventilation
* Patient refusal to participate

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2020-06-19 (Actual); Primary Completion 2021-11-18 (Actual); Study Completion 2021-11-18 (Actual)

PRIMARY OUTCOMES:
Time to spontaneous eye opening | At the end of surgery
  The interval from the cessation of anesthetics to spontaneous eye opening
Rate of in-hospital postoperative pulmonary complications | Within 30 days after surgery
  This includes atelectasis, pleural effusion, pneumonia, empyema, pulmonary embolism, re-operation, and respiratory failure. The diagnosis of atelectasis and pleural effusion will be made based on routinely performed chest radiographs on postoperative days 1 and 3. Pneumonia will be diagnosed if a patient presents with fever, leukocytosis and new infiltrates on chest radiography. Pleural empyema and pulmonary embolism will be confirmed by spiral computed tomography scan. Respiratory failure is defined as described in the protocol.

SECONDARY OUTCOMES:
Time to tracheal extubation | At the end of surgery
  The interval from the cessation of anesthetics to tracheal extubation
Time to orientation in time and place | At the end of surgery
  The interval from the cessation of anesthetics to orientation in time and place
Time to leave operating room | At the end of surgery
  The interval from the cessation of anesthetics to leave operating room
Rate of emergence agitation | During the recovery from anesthesia
  Richmond Agitation-Sedation Scale will be used to evaluate the level of agitation and sedation promptly after extubation. This is defined as +4 combative, +3 very agitated, +2 agitated, +1 restless, 0 alert and calm, -1 drowsy, -2 light sedation, -3 moderate sedation, -4 deep sedation, and -5 unarousable.
Rate of postoperative delirium | 30 minutes after tracheal extubation
  Events of delirium will be evaluated using the Confusion Assessment Method at the postanesthetic care unit.
Rate of intraoperative recall or awareness | One day after surgery
  As titled
Arterial partial pressure of oxygen (PaO2) / fraction of inspired oxygen (FiO2) | After induction of anesthesia and at the end of surgery
  The relative change of PaO2/FiO2 values after induction of anesthesia and at the end of surgery
Rate of cardiac complications | Within 30 days after surgery
  Myocardial infarction diagnosed by electrocardiogram and troponin T serum concentration; newly developed atrial fibrillation.
Rate of hypotensive episodes | Within 30 days after surgery
  This is defined as a decrease in mean arterial pressure > 20% for more than 15 min requiring vasopressors.
Rate of newly developed stroke | Within 30 days after surgery
  This will be based on the finding of imaging tests.
Length of hospital stay | Within 30 days after surgery
  As titled

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Hsuan Tai, M.D., M.Sc., Principal Investigator — Shuang-Ho Hospital, Taipei Medical University, New Taipei City, Taiwan
Locations (1):
- Shuang Ho Hospital, Taipei Medical University, Taipei, Taiwan

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-26): https://cdn.clinicaltrials.gov/large-docs/28/NCT04414228/Prot_SAP_000.pdf